CLINICAL TRIAL: NCT05094128
Title: Effectiveness of Upadacitinib in Patients With Axial Spondyloarthritis Suffering From Typical Disease Activity and Pain in a Real-World Setting
Brief Title: A Study to Assess Disease Activity in Adult Participants With Axial Spondyloarthritis Who Receive Upadacitinib in a Real-world Setting
Acronym: UpSPINE
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P21-007
Record Dates: First submitted 2021-10-20; First posted 2021-10-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Axial Spondylarthritis (r-axSpA)
Keywords: Axial Spondylarthritis (axSpA); Upadacitinib; RINVOQ
MeSH Terms: interventions — upadacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Upadacitinib.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Tablet; Oral
  Other Names: RINVOQ

SUMMARY:
Axial spondyloarthritis (axSpA) is an immune-mediated inflammatory disease primarily affecting the axial skeleton. The most frequent axSpA symptom is chronic, often inflammatory back pain that might be difficult to distinguish from other causes of chronic back pain. Many participants report persistent pain, including back pain, which impacts disease activity and and impairs quality of life while evoking typical disease burden such as sleep disturbance, social isolation, loss of productivity, as well as anxiety and depression. This study will assess the real-world effectiveness of upadacitinib on early and sustained disease control, and the association between pain and clinical/patient-reported outcomes in axSpA participants.

Upadacitinib is being developed for the treatment of axSpA. Approximately 352 adult participants with active axSpA will be enrolled in Germany.

Participants will receive oral upadacitinib tablets as prescribed by the physician prior to enrolling in this study in accordance with the terms of the local marketing authorization and professional and reimbursement guidelines with regards to dose, population and indication. The overall duration of the study is approximately 52 weeks.

There may be a higher burden for participants in this study compared to usual standard of care due to study procedures. Participants will attend regular visits per routine clinical practice. The effect of the treatment will be checked by medical assessments, checking for side effects, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of axSpA upon physician's judgement.
* Physician decision on participant treatment with upadacitinib must have been reached prior to and independently of recruitment in the study.
* Upadacitinib prescribed in accordance with the local label.

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor (including but not limited to upadacitinib, tofacitinib, baricitinib, and filgotinib).
* Participants with primary fibromyalgia (upon physician´s judgement)
* Participation in a clinical trial of an investigational drug, concurrently or within the last 30 days or five half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study.
* Participants who cannot be treated with upadacitinib according to the applicable local label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with axial spondylarthritis (axSpA) who have been prescribed upadacitinib in the course of routine practice according to relevant approved licenses.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Ankylosing Spondylitis Disease Activity Score Low Disease Activity (ASDAS LDA [< 2.1]) | Week 24
  The ASDAS combines the following 5 disease activity variables: back pain (BASDAI Question 2 NRS score 0 - 10), peripheral pain/swelling (BASDAI Question 3 NRS score 0 - 10), duration of morning stiffness (BASDAI Question 6 NRS score 0 - 10), PtGA, and high-sensitivity c reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR). Low disease is defined as an ASDAS < 2.1.
Percentage of Participants Achieving ASDAS LDA (< 2.1) (i.e., Maintenance of Response) | Up to Week 52
  The ASDAS combines the following 5 disease activity variables: back pain (BASDAI Question 2 NRS score 0 - 10), peripheral pain/swelling (BASDAI Question 3 NRS score 0 - 10), duration of morning stiffness (BASDAI Question 6 NRS score 0 - 10), PtGA, and high-sensitivity c reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR). Low disease is defined as an ASDAS < 2.1. Maintenance of response is defined as those achieving LDA at Week 24 and Week 52.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Assessment of Spondyloarthritis International Society Health Index (ASAS-HI) Score of 40 | Up to Week 52
  The ASAS-HI has been developed to measure functioning and health in participants with SpA with the aim of defining and comparing the impact of the disease and health based on the biopsychosocial model of disease proposed by the International Classification of Functioning, Disability and Health (ICF).
Percentage of Participants Achieving Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score < 4 | Up to Week 52
  The BASDAI is a commonly used measure to define disease activity levels in axSpA participants. The overall BASDAI score ranges from 0 to 10, with higher scores indicating greater disease activity.
Percentage of Participants Achieving ASDAS Inactive Disease (ID [< 1.3]) | Up to Week 52
  The ASDAS combines the following 5 disease activity variables: back pain (BASDAI Question 2 NRS score 0 - 10), peripheral pain/swelling (BASDAI Question 3 NRS score 0 - 10), duration of morning stiffness (BASDAI Question 6 NRS score 0 - 10), PtGA, and high-sensitivity c reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR). Inactive disease is defined as an ASDAS < 1.3.
Percentage of Participants Achieving ASDAS LDA (< 2.1) | Up to Week 52
  The ASDAS is a composite index with proven validity and reliability to assess disease activity in axSpA participants, with LDA defined as a score < 2.1.
Change from Baseline in BASDAI | Up to Week 52
  The BASDAI is a commonly used measure to define disease activity levels in axSpA participants. The overall BASDAI score ranges from 0 to 10, with higher scores indicating greater disease activity.
Change from Baseline in BASDAI at Week 1-4 | Week 4
  The BASDAI is a commonly used measure to define disease activity levels in axSpA participants. The overall BASDAI score ranges from 0 to 10, with higher scores indicating greater disease activity.
Percentage of Participants with Resolution of Enthesitis (Leeds Enthesitis Index [LEI] = 0) for Participants with Baseline Enthesitis | Up to Week 52
  The LEI is a clinical index used to assess enthesitis. It consists of 3 bilateral sites: Achilles tendon insertions, medial femoral condyles, and lateral epicondyles of the humerus. Tenderness at each site is quantified on a dichotomous basis: 0 means nontender and 1 means tender.
Percentage of Participants with Resolution of Dactylitis for Participants with Baseline Dactylitis | Up to Week 52
  Presence of dactylitis (Yes/No) will be assessed by the physician.
Mean Change from Baseline in ASAS-HI | Up to Week 52
  The ASAS-HI has been developed to measure functioning and health in patients with SpA with the aim of defining and comparing the impact of the disease and health based on the biopsychosocial model of disease proposed by the ICF.
Percentage of Participants with ASAS-HI <= 4 | Up to Week 52
  The ASAS-HI has been developed to measure functioning and health in patients with SpA with the aim of defining and comparing the impact of the disease and health based on the biopsychosocial model of disease proposed by the ICF.
Mean Change from Baseline in Nocturnal Back Pain in Past 24 Hours | Up to Week 52
  Pain will be measured using a 0 - 10 numerical rating scale (NRS) for nocturnal back pain (0 = no pain and 10 = most severe pain).
Mean Change from Baseline in Total Back Pain in Past 24 Hours | Up to Week 52
  Pain will be measured using a 0 - 10 numerical rating scale (NRS) for nocturnal back pain (0 = no pain and 10 = most severe pain).
Mean Change from Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) | Up to Week 52
  The BASFI is a validated PRO instrument for use in the axSpA participant population. It consists of 10 items measured on a 0 to 10 NRS, which assesses the ability to perform activities known to be problematic to axSpA participants such as dressing, bending, reaching, turning, and climbing steps. The total scores range from 0 to 10 with higher scores indicating worse physical functioning in axSpA participants.
Mean Change from Baseline in Patient Health Questionnaire-4 (PHQ-4) | Up to Week 52
  The 4-item PHQ-4 is an ultra-brief self-report questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2). It is rated on a 4-point Likert-type scale. Its purpose is to allow for very brief and accurate measurement of depression and anxiety.
Percentage of Participants with Recurrence of Typical Extra-Musculoskeletal Manifestations (EMMs) | Up to Week 52
  Participants with recurrence of typical extra-musculoskeletal manifestations (EMMs.
Percentage of Participants with new onset of typical EMMs | Up to Week 52
  Participants with new onset of typical EMMs

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (72):
- Germany (72):
  - ACURA Rheumazentrum Baden-Bade /ID# 249751, Baden-Baden, Baden-Wurttemberg
  - Heilig, Heidelberg, DE /ID# 240492, Heidelberg, Baden-Wurttemberg
  - Rheumatologische Schwerpunktpraxis /ID# 245392, Stuttgart, Baden-Wurttemberg
  - Praxis Dr. Haas /ID# 242982, Tübingen, Baden-Wurttemberg
  - Praxis Dr. Rinaldi /ID# 242984, Ulm, Baden-Wurttemberg
  - Praxis K. Pagel /ID# 240490, Hoppegarten, Brandenburg
  - Rheumahaus Studien GbR, Potsdam, DE /ID# 245231, Potsdam, Brandenburg
  - Praxis Dr. Sabine Reckert /ID# 245142, Potsdam, Brandenburg
  - Fachpraxis fuer Rheumatologie und Osteologie /ID# 243358, Bruchhausen-Vilsen, Lower Saxony
  - Stille, Hanover, DE /ID# 252222, Hanover, Lower Saxony
  - Praxis. F. Bigdeli-Wilshusen /ID# 272904, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover /ID# 262814, Hanover, Lower Saxony
  - Rheumatologie Kassel /ID# 275998, Kassel, Lower Saxony
  - Krankenhaus Porz am Rhein /ID# 243765, Cologne, North Rhine-Westphalia
  - Rheumazentrum Ruhrgebiet /ID# 240460, Herne, North Rhine-Westphalia
  - Beyer, Kaiserslautern, DE /ID# 240444, Kaiserslautern, Rhineland-Palatinate
  - Krankenhaus der Barmherzigen Brüder Trier /ID# 240524, Trier, Rhineland-Palatinate
  - Praxis Bernd Mueller /ID# 240488, Homburg, Saarland
  - Rheumapraxis Dr. Prothmann /ID# 240671, Püttlingen, Saarland
  - Medizinischen Versorgungszentrums Agilomed /ID# 240481, Chemnitz, Saxony
  - Rheumatologisches Medizinisches Versorgungszentrum Dresden /ID# 240516, Dresden, Saxony
  - Hamann & Teich & Boche,Leipzig /ID# 240445, Leipzig, Saxony
  - Praxis internistische Rheumatologie /ID# 240515, Leipzig, Saxony
  - Praxis Dr. Liebhaber /ID# 240480, Halle, Saxony-Anhalt
  - Aurich & Sieburg, Magdeburg /ID# 240518, Magdeburg, Saxony-Anhalt
  - Rheumatologische Praxis Dr. Jochen Walter /ID# 250263, Rendsburg, Schleswig-Holstein
  - MVZ Ambulantes Rheumazentrum Erfurt /ID# 244448, Erfurt, Thuringia
  - Rheumapraxis Weimar /ID# 268387, Weimar, Thuringia
  - Kupka & Kupka, Altenburg, DE /ID# 240479, Altenburg
  - Marycz, Amberg, DE /ID# 240483, Amberg
  - Rheumapraxis am Webereck /ID# 240454, Augsburg
  - Praxis S. Bresgulewski /ID# 240662, Bad Bertrich
  - Kerckhoff Klinik /ID# 252219, Bad Nauheim
  - Rheumapraxis Berlin /ID# 242987, Berlin
  - Praxis Dr. med. Angela Seifert /ID# 245107, Berlin
  - Praxis Dr. Silke Zinke /ID# 240526, Berlin
  - Krankenhaus Waldfriede /ID# 268389, Berlin
  - Eisterhues, Braunschweig, DE /ID# 239438, Braunschweig
  - MVZ Herzogin Elisabeth Hospital /ID# 267983, Braunschweig
  - Dr. Walberer /ID# 249752, Burglengenfeld
  - Private Practice - Dr. Sebastian Schuh /ID# 240498, Coburg
  - Dres. Karger/Baerlecken /ID# 240442, Cologne
  - MVZ-Medizinisches Versorgungszentrum Daun GmbH /ID# 254839, Daun
  - Kreiskrankenhaus Demmin /ID# 240451, Demmin
  - Praxis Dilltal /ID# 240520, Ehringshausen
  - Private Practice - Dr. Daniel Bestler /ID# 251860, Erfurt
  - Michael Mueller, Freiberg, DE /ID# 240489, Freiberg
  - Praxis Dres. Sensse/Sensse /ID# 240517, Gifhorn
  - Private Practice - Dr. Hauke E. Heintz /ID# 254037, Hamburg
  - Dres. Weinhardt/Knobel/Doepfer /ID# 248195, Hamburg
  - Zentrum fuer Rheumatologie und Schmerzmedizin /ID# 244370, Hanover
  - Wernicke, Hohen Neuendorf, DE /ID# 250626, Hohen Neuendorf
  - Kremers, Juelich, DE /ID# 243357, Jülich
  - Dr. Bolze, Ludwigshafen, DE /ID# 251012, Ludwigshafen
  - Praxis Dr. Annekatrin Rossbach /ID# 240495, Mansfeld / Großörner
  - Harmuth, Marktredwitz, DE /ID# 240455, Marktredwitz
  - RHIO Forschungsinstitut /ID# 240525, Meerbusch
  - Prof-med-stud.de /ID# 240458, Munich
  - Rheumatologische Facharztpraxis /ID# 240477, Naumburg
  - Praxis Dr. med Thilo Klopsch /ID# 240461, Neubrandenburg
  - Praxis Hein & Gess /ID# 240456, Nienburg
  - MVZ für Rheumatologie Dr. M. Welcker /ID# 240521, Planegg
  - Baumann & Lang, Plauen, DE /ID# 244369, Plauen
  - Rheumazentrum Ratingen /ID# 240465, Ratingen
  - Melzer, Seesen, DE /ID# 240484, Seesen
  - Barmherzige Bruder MVZ Klinikum Straubing GmbH /ID# 240523, Straubing
  - Rheumathologie Ulm /ID# 240494, Ulm
  - Praxis F. Schattenberg /ID# 257646, Waren
  - Krankenhaus St. Josef /ID# 249747, Wuppertal
  - Praxis Barmen /ID# 240449, Wuppertal
  - Praxis Barmen /ID# 277515, Wuppertal
  - Fricke-Wagner, Zwickau, DE /ID# 240452, Zwickau

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/